CLINICAL TRIAL: NCT05718986
Title: Epidemiology of Familial B-cell Lymphoproliferative Disorders
Brief Title: Familial B-cell Lymphoproliferative Disorders
Acronym: Familial_LPD
Status: Not yet recruiting | Type: Observational
Sponsor: University of Haifa (Other)
Collaborators: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Geffen Kleinstern, Senior Lecturer, University of Haifa
Other Study IDs: FamilialLPD
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Lymphoproliferative Disorders; Premalignant; Monoclonal B-Cell Lymphocytosis; Chronic Lymphocytic Leukemia
Keywords: lymphoproliferative disorders; Chronic Lymphocytic Leukemia; Monoclonal B-cell Lymphocytosis
MeSH Terms: conditions — Lymphoproliferative Disorders; Precancerous Conditions; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Blood and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (15):
- Bnai Zion Medical Center: Bnai Zion Medical Center
  Interventions: Other: No intervention
- Tel Aviv Sourasky Medical Center - Ichilov Hospital: Tel Aviv Sourasky Medical Center - Ichilov Hospital
  Interventions: Other: No intervention
- Galil Medical Center: Galil Medical Center
  Interventions: Other: No intervention
- Ziv Medical Center: Ziv Medical Center
  Interventions: Other: No intervention
- Emek Medical Center: Emek Medical Center
  Interventions: Other: No intervention
- Beilinson Hospital: Beilinson Hospital
  Interventions: Other: No intervention
- Meir Medical Center: Meir Medical Center
  Interventions: Other: No intervention
- Kaplan Medical Center: Kaplan Medical Center
  Interventions: Other: No intervention
- Sheba Medical Center: Sheba Medical Center
  Interventions: Other: No intervention
- Rambam Medical Center: Rambam Medical Center
  Interventions: Other: No intervention
- Shaare Zdek Medical Center: Shaare Zdek Medical Center
  Interventions: Other: No intervention
- Hadassah Medical Center: Hadassah Medical Center
  Interventions: Other: No intervention
- Shamir Medical Center (Assaf Harofeh): Shamir Medical Center (Assaf Harofeh)
  Interventions: Other: No intervention
- Soroka Medical Center: Soroka Medical Center
  Interventions: Other: No intervention
- Assuta Ashdod Hospital: Assuta Ashdod Hospital
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study investigates families with at least two cases of B-cell lymphoproliferative disorders (LPD), and evaluates the prevalence of LPD in families, the relationship between medical history, genetic factors, and the risk of familial LPD, and various clinical outcomes for these families in a multiethnic population of Jews and Arabs in Israel.

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion criteria:

Patients must have LPD and must have a family history of LPD. LPD patients who signed an informed consent to participate in the study.

Criteria for the inclusion of relatives of patients:

Relatives must be related by blood to LPD patients or unrelated (for control group).

Relatives who signed an informed consent to participate in the study.

Exclusion Criteria:

* Pregnant women, special populations and those lacking judgment will not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Jewish and Arab LPD families with at least 2 family members with LPD.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of familial LPD in Israel | 5 years
Association between medical history and genetic variants and the risk of familial LPD | 5 years
Risk of clinical outcomes among familial LPD and family members | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Geffen Kleinstern, PhD, Principal Investigator — University of Haifa

IPD SHARING:
Plan to Share IPD: No